CLINICAL TRIAL: NCT00710385
Title: Reinforcing Effects of Intravenous Buprenorphine Versus Buprenorphine/Naloxone in Buprenorphine-maintained Intravenous Drug Users (P05207)
Brief Title: Abuse Liability of Suboxone Versus Subutex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 5518
Record Dates: First submitted 2008-06-11; First posted 2008-07-04 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Opioid-related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Heroin; Naloxone; Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Heroin (Active Comparator): Heroin 25 mg. Administered intravenously, while participants were under 2, 8 and 24 sublingual (SL) Bup maintenance conditions.
  Interventions: Drug: Heroin
- Naloxone (Active Comparator): Naloxone (NAL) .4 mg. Administered intravenously, while participants were under 2, 8 and 24 sublingual (SL) Bup maintenance conditions.
  Interventions: Drug: Naloxone
- Low Bup Dose (Experimental): Combined dosing groups of (4 mg and 8mg of Buprenorphine) for participants who administered a maximum of 8 mg of Bup during the qualification phase. Administered intravenously, while participants were under 2, 8 and 24 sublingual (SL) Bup maintenance conditions.
  Interventions: Drug: Low Bup Dose
- Low Bup/Nal Dose (Experimental): Combined dosing groups of (4/1 mg and 8/2mg of Buprenorphine + Naloxone) for participants who administered a maximum of 8 mg of Bup during the qualification phase. Administered intravenously, while participants were under 2, 8 and 24 sublingual (SL) Bup maintenance conditions.
  Interventions: Drug: Low Bup/Nal Dose
- High Bup Dose (Experimental): Combined dosing groups of (8mg and 16mg of Bup) for participants who administered a maximum of 16 mg of Bup during the qualification phase. Administered intravenously, while participants were under 2, 8 and 24 sublingual (SL) Bup maintenance conditions.
  Interventions: Drug: High Bup Dose
- High Bup/Nal Dose (Experimental): Combined dosing groups of (8/2mg and 16/4mg of Buprenorphine + Naloxone) for participants who administered a maximum of 16 mg of Bup during the qualification phase. Administered intravenously, while participants were under 2, 8 and 24 sublingual (SL) Bup maintenance conditions.
  Interventions: Drug: High Bup/Nal Dose
- Placebo (Placebo Comparator): Intravenous placebo (PCB) administration. Administered intravenously, while participants were under 2, 8 and 24 sublingual (SL) Bup maintenance conditions.
  Interventions: Drug: Placebo (PCB)

INTERVENTIONS:
Drug: Heroin — Heroin (25 mg)
  Other Names: Diacetylmorphine
  Arms: Heroin
Drug: Naloxone — .4 mg
  Other Names: Naloxone Hydrochloride (HCl)
  Arms: Naloxone
Drug: Low Bup Dose — 4 and 8 mg
  Other Names: Subutex
  Arms: Low Bup Dose
Drug: High Bup Dose — 8mg and 16 mg
  Other Names: Subutex
  Arms: High Bup Dose
Drug: Low Bup/Nal Dose — Buprenorphine/Naloxone 4/1 mg, 8/2 mg
  Other Names: Suboxone
  Arms: Low Bup/Nal Dose
Drug: High Bup/Nal Dose — Buprenorphine/Naloxone 8/2 mg, 16/4 mg
  Other Names: Suboxone
  Arms: High Bup/Nal Dose
Drug: Placebo (PCB) — Placebo control administration
  Other Names: 0 mg
  Arms: Placebo

SUMMARY:
The study is designed to compare the abuse liabilities of intravenous buprenorphine and buprenorphine/naloxone in individuals who are physically dependent on sublingual buprenorphine. We hypothesize that the abuse liability of buprenorphine/naloxone is lower than that of buprenorphine alone.

DETAILED DESCRIPTION:
Drug dependence is a major international public health problem of which opioid dependence, notably involving heroin, is a major component. Opioid dependence affects an estimated 13 million injection drug users (IDUs) worldwide. The high health service costs for the treatment of diseases related to non-medical drug use and the high cost to society of drug-related behavior have prompted researchers to seek new medications and treatment strategies for opioid dependence. Buprenorphine, a mu-opiate receptor partial agonist and kappa-opiate receptor antagonist, is one such new medication that has had a significant role in expanding access to effective opioid dependence treatment. It is available as Subutex (buprenorphine alone) or Suboxone (a combination of buprenorphine and naloxone). Although it is commonly believed that the abuse potential of buprenorphine is low, numerous countries have reported illicit diversion of buprenorphine and a growing population of buprenorphine abusers. Theoretically, Suboxone would have lower abuse potential. When used sublingually, as prescribed, the amount of naloxone absorbed is negligible. However, if a patient crushes the tablet and attempts to inject or sniff the medication, the naloxone will become effective as an opioid antagonist and may precipitate withdrawal signs and symptoms in individuals dependent on full opioid agonists and/or attenuate the euphoric effects of the buprenorphine that is also contained in the medication. To date, few laboratory studies have evaluated the abuse liability of buprenorphine in humans using a drug self-administration protocol. We are proposing to evaluate the abuse potential of intravenous (IV) buprenorphine compared to IV buprenorphine/naloxone in buprenorphine-maintained injection drug users (IDUs), incorporating self-administration procedures with other measures of opioid effects. The proposed study will investigate the conditions that affect the self-administration of IV buprenorphine by buprenorphine abusers. The primary aim of the study is to compare the reinforcing effects of IV buprenorphine and IV buprenorphine/naloxone in IDUs maintained on different doses of sublingual buprenorphine (2, 8, and 24 mg/day). Secondary aims of the study are to compare the subjective, performance and physiological effects of IV buprenorphine and IV buprenorphine/naloxone. IV-administered placebo (saline), naloxone alone, and heroin alone will be tested as neutral, negative, and positive control conditions, respectively. Participants (N=12 completers) will reside on an inpatient unit (the General Clinical Research Unit, GCRU) during a 7 to 8-week study. This research will provide useful information for clinicians treating opioid dependent individuals with buprenorphine, and importantly, will provide information about the abuse potential and effects of buprenorphine on multiple measures of human functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual (DSM) IV criteria for heroin dependence
* No major mood, psychotic, or anxiety disorder
* Physically healthy
* Able to perform study procedures
* 21-45 years of age
* Normal body weight
* Current use of i.v. opioids in amounts and/or frequencies that meet or exceed those used in the proposed study (1-2 bags of heroin per occasion at least twice per day)
* Self-administer at least 4 mg i.v. buprenorphine above placebo levels during the dose run up phase

Exclusion Criteria:

* DSM IV criteria for dependence on drugs other than opioids, nicotine or caffeine
* Participants requesting treatment
* Participants on parole or probation
* Pregnancy or lactation
* Birth, miscarriage or abortion within 6 months
* Current or recent history of significant violent behavior
* Current major Axis I psychopathology, other than opioid dependence (e.g., mood disorder with functional impairment or suicide risk, schizophrenia), that might interfere with ability to participate in the study
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal
* Significant suicide risk
* Current chronic pain
* Sensitivity, allergy, or contraindication to opioids
* Current or recent (past 30 days) physical dependence on or treatment with methadone, buprenorphine, or the buprenorphine/naloxone combination

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, PhD, Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute/Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data have been published in a peer-reviewed journal.

REFERENCES:
- [Result] Comer SD, Sullivan MA, Vosburg SK, Manubay J, Amass L, Cooper ZD, Saccone P, Kleber HD. Abuse liability of intravenous buprenorphine/naloxone and buprenorphine alone in buprenorphine-maintained intravenous heroin abusers. Addiction. 2010 Apr;105(4):709-18. doi: 10.1111/j.1360-0443.2009.02843.x. PMID 20403021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment dates: September 10, 2007 - August 13, 2008 Location: Medical clinic
Groups:
- Intravenous Challenge Doses: This study employs a within-subjects design, all participants experienced all 7 intravenous challenge doses. The challenge doses were administered under 3 sublingual buprenorphine maintenance conditions. The data presented were collapsed across the 3 sublingual groups.
Period: Overall Study
Arm/Group | Intravenous Challenge Doses
Started | 17 (19 participants signed consent for the study 2 withdrew before any study procedures were initiated.)
Completed | 12
Not Completed | 5
Not completed — Did not qualify | 1
Not completed — Withdrawal by Subject | 1
Not completed — Undisclosed back pain | 1
Not completed — Physician Decision | 1
Not completed — Undisclosed excessive methadone use | 1

BASELINE CHARACTERISTICS:
Groups:
- Challenge Doses: This study employs a within-subjects design, all participant experience all challenge doses.
Arm/Group | Challenge Doses
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — verbal report verified by ID
  Participants
    <=18 years | 0
    Between 18 and 65 years | 12
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Drug's Breakpoint
Description: Measure of a drug's reinforcing effects. The "Breakpoint" is the point at which the participant stop performing an operant task (clicks on a mouse) in order to received the drug. Therefore, the reported breakpoint is the total amount of work the participant was willing to perform to receive the dose being tested
Time Frame: Single measurement taken following each of the 7 IV experimental doses
Population: Heroin users, not seeking treatment
Measure: Mean (Standard Deviation); unit: number of clicks on a mouse
Groups:
- Heroin: Intravenous heroin 25 mg
- Naloxone: Intravenous Naloxone HCl
- Low Bup Dose: Lower doses of intravenous buprenorphine alone.
- High Bup Dose: Higher doses of intravenous buprenorphine
- Lower Bup/Nal Dose: Lower doses of intravenous buprenorphine + naloxone.
- High Bup/Nal Dose: Higher doses of intravenous buprenorphine +naloxone
- Placebo: Control intravenous placebo drug administration.
Arm/Group | Heroin | Naloxone | Low Bup Dose | High Bup Dose | Lower Bup/Nal Dose | High Bup/Nal Dose | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
number of clicks on a mouse | 1200 (200) | 10 (10) | 1100 (180) | 1200 (190) | 300 (100) | 750 (175) | 0 (0)

2. Secondary Outcome: Drug "Liking"
Description: Participant's subjective ratings of how much they "Like" the dose they just received on a scale of 0 -100.
Time Frame: Peak (highest) rating obtained following drug administration throughout the entire 3 hr session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Heroin | Naloxone | Low Bup Dose | High Bup Dose | Lower Bup/Nal Dose | High Bup/Nal Dose | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
units on a scale | 41.5 (5) | 3 (2.7) | 29.8 (4) | 42.5 (5) | 10.5 (2.4) | 27 (4) | 1 (.6)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for daily throughout the study.
Description: An adverse event (AE) was defined as any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. A serious adverse event is any AE that was: Fatal, Life-threatening, Required or prolonged inpatient stay, Resulted in persistent or significant disability or incapacity.
Groups:
- Combined for All Study Conditions: This study employed a within-subjects design, all participants experienced all study conditions.
Arm/Group | Combined for All Study Conditions
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 4/17
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined for All Study Conditions (N=17)
urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1)
dizziness (Injury, poisoning and procedural complications) | 1 (1)
chest discomfort (Injury, poisoning and procedural complications) | 1 (1)
Mild Opioid Withdrawal (Injury, poisoning and procedural complications) | 3 (3)

LIMITATIONS AND CAVEATS:
The stringent criteria for enrollment, qualification and retention in this trial were highly selective for a certain subpopulation of opioid-dependent individuals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No